CLINICAL TRIAL: NCT05410522
Title: Effect of an Electrostimulation Program in Lung Transplant Recipients During Their Stay in the Intensive Critical Care Unit. Experimental Study
Brief Title: Electrostimulation Program for Lung Transplant Recipients in the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CuidReaTxLung01
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental lung transplant (Experimental): The training time will be 30 minutes in the morning and 30 minutes in the afternoon with a total daily work time of 60 minutes. The frequency of work will be different in each session, seeking in the morning routine a vascularization and improvement of muscle trophism and in the afternoon an aerobic endurance, activation of the working capacity of the tonic muscles to improve the stabilizing muscles and postural fitness.
  Interventions: Device: EMS Program
- Control lung transplant (No Intervention): Electro stimulation therapy will not be performed.

INTERVENTIONS:
Device: EMS Program — Lower limb electrostimulation therapy is scheduled for lung transplant patients. The therapy consists in the application of 2 daily 30-minute sessions that begin in the first 48 hours post-transplantation and are maintained daily until discharge from the hospital.
  Arms: Experimental lung transplant

SUMMARY:
This study aims to evaluate rectus femoris muscle mass in lung transplant recipients and the effect of a training program during ICU admission based on the use of electrical muscle stimulation (EMS)

DETAILED DESCRIPTION:
Lung transplantation is so far the only viable therapy for those individuals with a life-threatening chronic respiratory individuals with a chronic respiratory problem that compromises their life in a period of less than two years and the therapeutic options have been exhausted.

The investigators are dealing with individuals with a prolonged disease process, characterized mainly by the reduction of their respiratory capacities, which has a great impact on the basic activities of daily living.

Pulmonary involvement conditions the mobility of the individual, limiting physical activity and leading to episodes of dyspnea.

The aerobic capacity of the patient is very impaired before the transplant, although after the transplant, it continues in levels below normal for their age . This, resulting in episodes of dyspnea impacts on the extraction and utilization of muscular oxygen , which reduces mobility periods.

Limitations in physical activity and even mobility prior to physical activity and even mobility limitations prior to transplantation lead these individuals to marked muscular deterioration, which has an impact on both the general physical and psychological levels.

The aim of this study is assessment of muscle status in transplant recipients in lung transplant recipients after application of EMS therapy in the ICU.The sample is divided into two groups, a control group that will not receive EMS therapy and a control group that receive it.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the lung transplant list according to the criteria of the Health System.
* Those who attend the rehabilitation consultation of the hospital under study to undergo treatment prior to transplantation.
* They must receive the graft at the hospital under study and be admitted to the resuscitation unit at the same center for post-surgical follow-up.

Exclusion Criteria:

* Those who are rejected from the transplant list or deceased before the implant is performed.
* Lack of follow-up by the rehabilitation consultation.
* Are receiving treatment with muscle relaxants after admission to the ICU.
* Present skin alterations incompatible with EMS.
* Contraindications to perform the transplant proposed according to the criteria of the Health System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Variation of muscle mass in the quadriceps | Up to 6 months prior to transplantation, within 24 hours of admission and every seven days and/or until discharge from the ICU (up to 14 days).
  The quadriceps muscle mass of the lung transplant recipient will be measured prior to transplantation and will be monitored in the first 24 hours post-transplant and every 7 days from admission until hospital discharge.

SECONDARY OUTCOMES:
Mobility assessment according to ICU-Mobility scale (IMS) | Each day in the morning and afternoon, until discharge from ICU (up to 14 days).
  Ability to move during ICU admission. IMS is a scale containing 10 items ranging from 0 (no mobility at all) to 10 (walks unaided), which some authors have categorized binary (< 4 passive/active mobilization in bed and ≥ 4 active mobilization out of bed).
Leg strength according to Chair and Stand test | Up to 6 months prior to transplantation and at ICU discharge (up to 14 days)
  Leg strength assessment before transplantation and at discharge from ICU (up to 14 days), using Chair and Stand test

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Díaz-Teruel, MsD, Principal Investigator — Hospital Universitario 12 de Octubre; Ignacio Zaragoza-García, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Brandt J, Spruit MA, Hansen D, Franssen FM, Derave W, Sillen MJ, Burtin C. Changes in lower limb muscle function and muscle mass following exercise-based interventions in patients with chronic obstructive pulmonary disease: A review of the English-language literature. Chron Respir Dis. 2018 May;15(2):182-219. doi: 10.1177/1479972317709642. Epub 2017 Jun 5. PMID 28580854
- [Result] Shah S, Darekar B, Salvi S, Kowale A. Quadriceps strength in patients with chronic obstructive pulmonary disease. Lung India. 2019 Sep-Oct;36(5):417-421. doi: 10.4103/lungindia.lungindia_27_19. PMID 31464214
- [Result] Maury G, Langer D, Verleden G, Dupont L, Gosselink R, Decramer M, Troosters T. Skeletal muscle force and functional exercise tolerance before and after lung transplantation: a cohort study. Am J Transplant. 2008 Jun;8(6):1275-81. doi: 10.1111/j.1600-6143.2008.02209.x. Epub 2008 Apr 29. PMID 18444941
- [Result] Zhang L, Hu W, Cai Z, Liu J, Wu J, Deng Y, Yu K, Chen X, Zhu L, Ma J, Qin Y. Early mobilization of critically ill patients in the intensive care unit: A systematic review and meta-analysis. PLoS One. 2019 Oct 3;14(10):e0223185. doi: 10.1371/journal.pone.0223185. eCollection 2019. PMID 31581205
- [Result] Janaudis-Ferreira T, Mathur S, Deliva R, Howes N, Patterson C, Rakel A, So S, Wickerson L, White M, Avitzur Y, Johnston O, Heywood N, Singh S, Holdsworth S. Exercise for Solid Organ Transplant Candidates and Recipients: A Joint Position Statement of the Canadian Society of Transplantation and CAN-RESTORE. Transplantation. 2019 Sep;103(9):e220-e238. doi: 10.1097/TP.0000000000002806. PMID 31461743